CLINICAL TRIAL: NCT02963077
Title: A Phase I, Double-Blind Single and Multiple Ascending Dose Study to Assess Safety and Pharmacokinetics of A4250 as Monotherapy, and in Combination With Colonic Release Cholestyramine (A3384) or Commercially Available Cholestyramine (Questran™) in Healthy Subjects
Brief Title: A Safety and Pharmakokinetic Study of A4250 Alone or in Combination With A3384
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Albireo (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A4250-001; 2013-001175-21 (EudraCT Number)
Record Dates: First submitted 2016-11-01; First posted 2016-11-15 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Orphan Cholestatic Liver Diseases; Primary Biliary Cirrhosis; Progressive Familial Intrahepatic Cholestasis; Alagille Syndrome
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Cholestasis, progressive familial intrahepatic 1; Alagille Syndrome | interventions — Cholestyramine Resin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (24):
- Cohort 1 SAD - 0.1 mg A4250 (Experimental): Dose: 0.1 mg of A4250. Sentinel dosing was used (2 sub-cohorts dosed a minimum of 24 h apart).
  Interventions: Drug: A4250
- Cohort 2 SAD - 0.3 mg A4250 (Experimental): Dose: 0.3 mg of A4250.
  Interventions: Drug: A4250
- Cohort 3 SAD - 1 mg A4250 (Experimental): Dose: 1 mg A4250.
  Interventions: Drug: A4250
- Cohort 4 SAD - 3 mg A4250 (Experimental): Dose: 3 mg A4250.
  Interventions: Drug: A4250
- Cohort 5 SAD - 10 mg A4250 (Experimental): Dose: 10 mg A4250.
  Interventions: Drug: A4250
- Cohort 1 SAD placebo (Placebo Comparator): Dose: 0.1 mg of A4250 matching placebo. Sentinel dosing was used (2 sub-cohorts dosed a minimum of 24 h apart).
  Interventions: Drug: Placebo
- Cohort 2 SAD placebo (Placebo Comparator): Dose: 0.3 mg A4250 matching placebo.
  Interventions: Drug: Placebo
- Cohort 3 SAD placebo (Placebo Comparator): Dose: 1 mg A4250 matching placebo.
  Interventions: Drug: Placebo
- Cohort 4 SAD placebo (Placebo Comparator): Dose: 3 mg A4250 matching placebo.
  Interventions: Drug: Placebo
- Cohort 5 SAD placebo (Placebo Comparator): Dose: 10 mg A4250 matching placebo.
  Interventions: Drug: Placebo
- Cohort 1 MAD - 1 mg A4250 qd (Experimental): Dose: 1 mg A4250 qd for 7 days.
  Interventions: Drug: A4250
- Cohort 1 MAD placebo (Placebo Comparator): Dose: 1 mg A4250 matching placebo qd for 7 days.
  Interventions: Drug: Placebo
- Cohort 2 MAD - 3 mg A4250 (Experimental): Dose: 3 mg A4250 qd for 7 days
  Interventions: Drug: A4250
- Cohort 2 MAD placebo (Placebo Comparator): Dose: 3 mg A4250 matching placebo qd for 7 days.
  Interventions: Drug: Placebo
- Cohort 3 MAD - 1.5 mg A4250 b.i.d for 7 days. (Experimental): Dose: 1.5 mg A4250 b.i.d. for 7 days.
  Interventions: Drug: A4250
- Cohort 3 MAD placebo (Placebo Comparator): Dose: 1.5 A4250 matching placebo b.i.d for 7 days.
  Interventions: Drug: Placebo
- Cohort 4 MAD - 3 mg A4250 qd + 1 mg Questran b.i.d (Experimental): Dose: 3 mg A4250 qd + 1 mg Questran b.i.d for 7 days.
  Interventions: Drug: A4250; Drug: Questran
- Cohort 4 MAD A4250 placebo + 1 mg Questran b.i.d (Active Comparator): Dose: 3 mg A4250 matching placebo + 1 mg Questran b.i.d for 7 days.
  Interventions: Drug: Questran; Drug: Placebo
- Cohort 5 MAD - 3 mg A4250 qd + 1 g CRC b.i.d (Experimental): Dose: 3 mg A4250 qd + 1 g CRC b.i.d for 7 days.
  Interventions: Drug: A4250; Drug: CRC (A3384)
- Cohort 5 MAD A4250 placebo + CRC placebo (Placebo Comparator): Dose: 3 mg A4250 matching placebo qd + 1 g CRC placebo b.i.d for 7 days
  Interventions: Drug: Placebo
- Cohort 6 MAD - 1 g CRC (Active Comparator): Dose: 1 g CRC b.i.d
  Interventions: Drug: CRC (A3384)
- Cohort 6 MAD CRC placebo (Placebo Comparator): Dose: 1 g CRC matching placebo b.i.d.
  Interventions: Drug: Placebo
- Cohort 7 MAD - 3 mg A4250 qd + 1 g CRC b.i.d (Experimental): Dose: 3 mg A4250 qd + 1 g CRC b.i.d
  Interventions: Drug: A4250; Drug: CRC (A3384)
- Cohort 7 MAD A4250 placebo + CRC placebo (Placebo Comparator): Dose: 3 mg A4250 matching placebo qd + 1 g CRC matching placebo b.i.d.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: A4250
  Arms: Cohort 1 MAD - 1 mg A4250 qd; Cohort 1 SAD - 0.1 mg A4250; Cohort 2 MAD - 3 mg A4250; Cohort 2 SAD - 0.3 mg A4250; Cohort 3 MAD - 1.5 mg A4250 b.i.d for 7 days.; Cohort 3 SAD - 1 mg A4250; Cohort 4 MAD - 3 mg A4250 qd + 1 mg Questran b.i.d; Cohort 4 SAD - 3 mg A4250; Cohort 5 MAD - 3 mg A4250 qd + 1 g CRC b.i.d; Cohort 5 SAD - 10 mg A4250; Cohort 7 MAD - 3 mg A4250 qd + 1 g CRC b.i.d
Drug: CRC (A3384)
  Arms: Cohort 5 MAD - 3 mg A4250 qd + 1 g CRC b.i.d; Cohort 6 MAD - 1 g CRC; Cohort 7 MAD - 3 mg A4250 qd + 1 g CRC b.i.d
Drug: Questran
  Arms: Cohort 4 MAD - 3 mg A4250 qd + 1 mg Questran b.i.d; Cohort 4 MAD A4250 placebo + 1 mg Questran b.i.d
Drug: Placebo
  Arms: Cohort 1 MAD placebo; Cohort 1 SAD placebo; Cohort 2 MAD placebo; Cohort 2 SAD placebo; Cohort 3 MAD placebo; Cohort 3 SAD placebo; Cohort 4 MAD A4250 placebo + 1 mg Questran b.i.d; Cohort 4 SAD placebo; Cohort 5 MAD A4250 placebo + CRC placebo; Cohort 5 SAD placebo; Cohort 6 MAD CRC placebo; Cohort 7 MAD A4250 placebo + CRC placebo

SUMMARY:
The primary objectives of the study are to evaluate the safety, tolerability and pharmacokinetics of A4250 after single or multiple oral doses in healthy subjects. In addition, will evaluate A4250 in combination with cholestyramine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or non-pregnant, non-lactating healthy females
2. BMI of 18 to 32 kg/m2 or, if outside the range, considered not clinically significant by the investigator
3. Willing and able to communicate and participate in the whole study
4. Provided written informed consent
5. Agreed to use an adequate method of contraception

Exclusion Criteria:

1. Had participated in a clinical research study within the previous 3 months
2. Were study site employees, or immediate family members of a study site or sponsor employee
3. Had previously been enrolled in this study
4. History of any drug or alcohol abuse in the past 2 years
5. Regular alcohol consumption, in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
6. Current smokers and those who had smoked within the last 12 months. A breath carbon monoxide (CO) reading of greater than 10 ppm at screening
7. Females of childbearing potential who were pregnant or lactating (female subjects must have had a negative urine pregnancy test at admission)
8. Did not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
9. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator
10. Positive drugs of abuse test result
11. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
12. History of cardiovascular, renal, hepatic, chronic respiratory or GI disease as judged by the investigator
13. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients eg lactose or contraindications to cholestyramine/Questran
14. Presence or history of clinically significant allergy requiring treatment as per the judgement of the investigator Hayfever was allowed unless it was active
15. Donation or loss of greater than 400 mL of blood within the previous 3 months
16. Were taking, or had taken, any prescribed or over-the-counter drug (other than up to 4 g per day paracetamol, hormone replacement therapy [HRT] and hormonal contraception) or herbal remedies in the 14 days before IMP administration unless they were not considered to have interfered with the objectives of the study, as agreed by the PI and sponsor's medical monitor on a case by case basis
17. Failed to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Mean (± SD) Plasma Pharmacokinetic Concentrations of A4250 Following A Single Oral 10 mg A4250 Dose - Tmax | Pharmacokinetic blood samples were taken pre-dose, and post-dose at: 0.5 hour, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours and 24 hours
Mean (± SD) Plasma Pharmacokinetic Concentrations of A4250 Following a Single Oral 10 mg A4250 Dose - Cmax | Pharmacokinetic blood samples were taken pre-dose, and post-dose at: 0.5 hour, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours and 24 hours
Mean (± SD) Plasma Pharmacokinetic Concentrations of A4250 Following a Single Oral 10 mg A4250 Dose - AUC 0-t | Pharmacokinetic blood samples were taken pre-dose, and post-dose at: 0.5 hour, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours and 24 hours
Mean (SD) Change in FGF19 from Day 1 Pre-Dose to 4 h Post-Dose | Pharmacodynamic blood samples were taken pre-dose and at 4 hours and 24 hours post-dosing, and at follow-up (5-7 days after final dose).
Mean (SD) Change in FGF19 from Day 1 Pre-Dose to 24 h Post-Dose | Pharmacodynamic blood samples were taken pre-dose and at 4 hours and 24 hours post-dosing, and at follow-up (5-7 days after final dose).
Mean (SD) Change in C4 from Day 1 Pre-Dose to 4 h Post-Dose | Pharmacodynamic blood samples were taken pre-dose and at 4 hours and 24 hours post-dosing, and at follow-up (5-7 days after final dose).
Mean (SD) Change in C4 from Day 1 Pre-Dose to 24 h Post-Dose | Pharmacodynamic blood samples were taken pre-dose and at 4 hours and 24 hours post-dosing, and at follow-up (5-7 days after final dose).
Mean (SD) Changes in Total Bile Acids for A4250 4 h compared to pre-dose | Samples were taken pre-dose and post-dose at 4 hours and 24 hours.
Mean (SD) Changes in Total Bile Acids for A4250 24 h compared to pre-dose | Samples were taken pre-dose, and post-dose at 4 hours and 24 hours.
Geometric (geometric CV%) Mean for AUC(0-12) on Day 7 for plasma FGF19 | AUC(0-12) on Day 7 (only for Part II)
Geometric (geometric CV%) Mean for AUC(0-12) on Day 7 for plasma C4 | AUC(0-12) on Day 7 (only Part II)
Geometric (geometric CV%) Mean for AUC(0-12) on Day 7 for plasma Total Bile Acids | AUC(0-12) on Day 7 (only Part II)
Mean (SD) Changes in Faecel Total Bile Acids from Day 1 Pre-Dose on Day 7 at 24 h Post-dose | Change from Day 1 Pre-dose to Day 7 at 24 hours Post-dose
Mean (SD) Change in Faecal Total Bile Acids Excreted (ng) from Day 1 Pre-Dose on Day 7 Post-Dose | Change from Day 1 Pre-dose to Day 7 at 24 hours Post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen

IPD SHARING:
Plan to Share IPD: No